CLINICAL TRIAL: NCT04766125
Title: Psychological Factors in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AUPsych
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Conditions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard adverse event information (Other)
  Interventions: Behavioral: Adverse event information
- Elaborated adverse event information (Other)
  Interventions: Behavioral: Adverse event information

INTERVENTIONS:
Behavioral: Adverse event information — All patients have access to the standard material about adverse events related to the surgery. One arm will additionally receive elaborated adverse event information from a nurse and a surgeon

SUMMARY:
The study investigates the effect of adverse event information on adverse event occurrence in patients undergoing elective cardiac surgery in a two-armed, randomized study. One group will receive standard information about adverse events; the second group will receive a standardised elaboration of the standard information. Hypothesis: Elaborated information about adverse events will increase adverse event occurrence, mediated by expectations and anxiety, and moderated by coping style.

DETAILED DESCRIPTION:
If quality assessment indicates that the protocol was not followed adequately, participants will be excluded from data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 and older) undergoing elective cardiac surgery at the Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital

Exclusion Criteria:

* Patients who have previously had cardiac surgery
* Cardiac surgery with deep hypothermia (<32 degrees Celsius)
* Acute surgery
* Patients with psychiatric or neurological disease who are unable to collaborate with the study protocol
* Patients who do not speak/read Danish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Assessed on day four

SECONDARY OUTCOMES:
Number of adverse events | Assessed on day 30, 90, and 180
Intensity of experienced adverse events | Assessed on day four, 30, 90, and 180
Hospital readmission | Assessed on day 180
Occurrence of specific adverse events | Assessed on day four, 30, 90, and 180

CONTACTS AND LOCATIONS:
Overall Officials: Mette Sieg, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No